CLINICAL TRIAL: NCT04871893
Title: Safety and Effcacy Evaluation of CO2 Removal in Combination With Continuous Veno-Venous Hemodialysis/Hemodiafiltration Therapy (A Clinical Study in Patients With Combined Renal Failure and Hypercapnia Due to Acute Lung Failure in COVID-19 and Other Forms of Respiratory Insufficiency)
Brief Title: Safety and Efficacy Evaluation of CO2 Removal in Combination With Continuous Veno-Venous Hemodialysis/Hemodiafiltration Therapy
Acronym: multiECCO2R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: CERES GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRRT-CVVHD/HDF-01-D; CIV-21-03-035951 (Other: Unique identification number EUDAMED)
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Acute Lung Injury; Acute Kidney Injury; Hypercapnia; Covid19
Keywords: CO2 removal; Continuous Renal Replacement Therapy; blood-gas exchanger; CRRT; multiECCO2R
MeSH Terms: conditions — Acute Lung Injury; Acute Kidney Injury; Hypercapnia; COVID-19

STUDY DESIGN:
Intervention Model Description: Prospective, non-comparative, multi-centre, open-label, interventional PMCF study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with the blood-gas exchanger multiECCO2R for CO2 removal (Other): Treatment of patients suffering from hypercapnia due to acute lung failure and acute kidney injury (AKI). Patients will be treated up to 72 hours with CVVHD/HDF with a standard multiFiltrate blood line kit (multiFiltrate or multiFiltrate Pro). In order to perform an ECCO2R procedure during CVVHD/HDF treatment, the blood-gas exchanger multiECCO2R is inserted in a specifically designed blood line kit downstream of the hemodialyzer.
  Interventions: Device: multiECCO2R blood-gas exchanger

INTERVENTIONS:
Device: multiECCO2R blood-gas exchanger — Treatment with the blood-gas exchanger multiECCO2R for CO2 removal

SUMMARY:
Objective of the study is to assess the safety and efficacy of CO2 removal by the multiECCO2R (CO2 Removal System) on the multiFiltrate/multiFiltrate Pro in veno-venous extracorporeal circulation during continuous renal replacement therapy (CRRT) in patients presenting with hypercapnia due to acute lung failure and acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated by the investigator; and:

  1. if patient is able to give consent: by the study patient
  2. if patient is unable to give consent: by the legal representative or
  3. if an emergency situation is determined: by an independent consultant physician
* Minimum age of 18 years

Study-specific:

* Body weight greater than 40 kg
* Acute Kidney Injury (AKI) with clinical indication for CRRT
* Hypercapnia with indication for ECCO2R:

(paCO2 ≥ 55 mmHg at given best possible protective ventilation parameters: Guiding parameters: tidal volume = 6 ml/kg PBW, PEEP to be adjusted according to the FiO2 1, driving pressure < 15 cmH2O, max. inspiratory pressure < 30 cmH2O or TV<=5 ml/kg when max. inspiratory pressure< 30 cmH2O cannot be held)

* Vascular access and Shaldon catheter allowing blood flow of 100 ml/min to 500 ml/min
* Arterial line in place, allowing blood sampling
* Estimated life expectancy greater than 3 days

Exclusion Criteria:

* In case of female patients: pregnancy or lactation period (if patient is ≥ 55 years old or have been surgically sterilized, a negative pregnancy test is not required)
* Participation in an interventional clinical study during the preceding 72 hours
* Previous participation in the same study

Study-specific

* Severe ARDS (Berlin definition): PaO2/FiO2 < 100 mmHg
* Intracerebral haemorrhage
* Intracranial hypertension
* Acute myocardial infarction
* Hypersensitivity to heparin or known history of heparin induced thrombocytopenia (HIT Type II), if heparin is used as anticoagulant
* severe liver insufficiency or fulminant hepatic failure
* Uncontrolled bleeding and coagulation disorders, thrombocytopenia < 75000µL
* Liver cirrhosis CHILD Pugh Classification > A
* BMI > 40 kg/m²
* Decision to limit therapeutic interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical efficiency variables: Change of PaCO2 | 30 minutes after start of treatment
  Change of PaCO2 during the first 30 minutes of treatment (Blood-gas analysis (BGA))

SECONDARY OUTCOMES:
Technical efficiency variables: Change of pCO2 | 72 hours after start of treatment
  Change of pCO2 within the extracorporeal circuit by pre- and post- CO2-exchanger during the treatment (Blood-gas analysis (BGA))

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Müller, Prof. Dr., Study Director — Universitätsklinikum Regensburg, Klinik und Poliklinik für Innere Medizin; Matthias Lubnow, Dr. med., Principal Investigator — Universitätsklinikum Regensburg, Klinik und Poliklinik für Innere Medizin
Locations (6):
- Germany (6):
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Universitätsklinikum Regensburg Klinik und Poliklinik für Innere Medizin, Regensburg, Bavaria
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum Donaustauf, Donaustauf
  - Universitätsklinikum Hamburg, Hamburg
  - Klinikum Herford, Herford